CLINICAL TRIAL: NCT03479190
Title: A Double Blind Randomised Control Trial Investigating the Efficacy of Platelet Rich Plasma Versus Placebo for the Treatment of Greater Trochanteric Pain Syndrome (HiPPO Trial)
Brief Title: Platelet Rich Plasma Versus Placebo for the Treatment of Greater Trochanteric Pain Syndrome (HiPPO Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mohammed Ali, Research Fellow, Northumbria Healthcare NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRAS 198415
Record Dates: First submitted 2018-03-13; First posted 2018-03-27 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Greater Trochanteric Pain Syndrome

STUDY DESIGN:
Intervention Model Description: The trial will be a two arm single centre double blind randomised control trial. The study will include a two-way comparison between PRP and placebo normal saline injections for treating GTPS. Participants will be reviewed at baseline, 3, 6 and 12 with patient reported outcome measures (PROM) completed at each of these reviews.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma (Active Comparator): ultrasound guided injection of Platelet rich plasma
  Interventions: Procedure: ultrasound guided injection of Platelet rich plasma
- Normal saline (Placebo Comparator): ultrasound guided injection of Normal saline
  Interventions: Procedure: ultrasound guided injection of Normal Saline

INTERVENTIONS:
Procedure: ultrasound guided injection of Platelet rich plasma — Platelet rich plasma (PRP) injection into trochanteric area under ultrasound guidance
  Arms: Platelet rich plasma
Procedure: ultrasound guided injection of Normal Saline — ultrasound guided injection of Normal Salineinto trochanteric area under ultrasound guidance
  Arms: Normal saline

SUMMARY:
Greater Trochanteric Pain Syndrome (GTPS), also known as Trochanteric Bursitis, is a painful condition predominantly affecting middle aged women. It is characterised by pain in the lateral hip exacerbated by movement and lying on the affected side. GTPS encompasses different conditions including gluteus medius/minimus tendinopathy and bursal inflammation. The treatment for this condition begins with conservative treatments of analgesia and physiotherapy, which normally results in a resolution of symptoms. If this fails then steroid injections have been shown to be effective. If this is not successful patients are offered surgery. Steroid injections however may only be effective in the short term and sometimes patients require repeat injections. Platelet rich plasma (PRP) is plasma taken from the blood of the patient that has been treated so that it has a higher than usual concentration of platelets in it. It has been postulated to promote healing in damaged or inflamed tissues. Platelets contain a variety of growth factors, which are involved in healing. It has been used in a variety of orthopaedic conditions such as lateral elbow epicondylitis, patellar tendonitis, rotator cuff pathology and planter fasciitis. Studies have shown varying effects of PRP in these conditions with most promise in plantar fasciitis and patellar tendonitis. These conditions are similar to GTPS. A recent review of treatments for GTPS concluded that more research into PRP efficacy in GTPS is required. We hypothesise that PRP is effective in treating GTPS in patients who have not responded to conservative management (analgesia and physiotherapy). This is an area that lacks research and could be valuable to those suffering from GTPS. Further study is required as PRP could be used as instead of steroid injections or if steroid treatments have failed and this could prevent patients from suffering further or needing surgery.

The investigators propose a randomised control trial comparing a normal saline injection with a PRP injection in patients with GTPS, diagnosed by MRI scan, who have not responded to conservative treatments. Patients will receive either PRP or normal saline under ultrasound guidance by a consultant rheumatologist. Sample size calculation has shown that the investigators will need to recruit a total of 100 patients who will be randomised into either arm (50 in each arm). The recruitment period will last 2 years with the whole trial aiming to finish in 4 years from the proposed start date. Neither patients or the study team members assessing the outcomes will know which treatment the patient received. Patients will be followed up at 3, 6 and 12 months. The primary outcome measure will be a patient reported outcome measure (PROM) i-HOT12 (international hip outcome tool) which is a valid and reliable scoring system that assesses patient's ability to return to an active lifestyle through obtaining subjective measures of symptoms, as well as determining emotional and social health status.

This will be alongside secondary outcome measures Visual Analogue Pain Score, Modified Harris Hip Score and EQ-5D collected. The proposal was discussed with a group of patients who previously had treatment with Platelet Rich Plasma (PRP) injection for hip pain. A discussion was had with regards the setup of a study and they were enthusiastic about this. A patient information sheet was shown to them and modified as per their comments. Their advice was obtained with regards the setup of this study, the randomisation into placebo arm, followup frequency and the outcome measures. In particular, patients suggested that if placebo was not working then a switch over to treatment arm should be discussed sooner than the initially planned one year. This has been taken into account and six month has been agreed. The proposal was also discussed in the NRES committee who are satisfied with the proposal. Ethical approval has been granted and the study is registered with Health Research Authority England.

DETAILED DESCRIPTION:
1. What is the problem being addressed? Greater trochanteric pain syndrome (GTPS), also known as trochanteric bursitis, is a painful condition characterised by pain around the greater trochanter usually affecting middle aged women (1). It was first described, as trochanteric bursitis in 1958 (2). Further details on the clinical symptoms published in 1978 as pain over the greater trochanter on walking, squatting or climbing stairs and pain on lying on the affected side or when crossing one's legs (3). Little described tenderness over the greater trochanter over the insertion of the gluteus tendons. GTPS was a term used by Karpinski et al 1985 instead of trochanteric bursitis as patients did not exhibit typical bursitis signs of swelling, heat, crepitus or fluctuation (4). This notion has been supported by other studies (5) including a study performed by Bird et al 2001 evaluated 24 patients using MRI with the clinical picture of GTPS and found that majority of them had gluteus medius tendon pathology with only 2 patients with trochanteric bursal inflammation (1). Hence, GTPS instead of trochanteric bursitis appears to be the more accurate way of described the clinical condition which seems to have multiple facets in its pathology.
2. Why is the research important? Greater trochanteric pain syndrome (GTPS) is one of the most common causes of lateral hip pain in adults and can be a painful and debilitating condition which as a last resort requires surgery especially if it does not respond to conservative treatments. The best estimates of prevalence are from a large, community-based study with over 3000 adults aged 50 to 70 years, in which unilateral GTPS was present in 15 percent of women and 6.6 percent of men. Bilateral GTPS was reported in 8.5 and 1.9 percent of women and men, respectively. The usual age at presentation is over 50 years, and the female to male ratio is approximately 4:1. It can be associated with low back pain in 20-35%. Bilateral GTPS in particular is associated with higher 20-meter walk time and chair stand time. It can lead to substantial limitation of activity and poor quality of life. It is therefore important to look at appropriate treatment options that will lead to quicker and more long-lasting recovery.

   Currently the treatment ladder for GTPS consists of conservative measures such as physiotherapy and NSAIDs. The majority of patients will settle with conservative management however if this fails then more invasive treatment options include shockwave therapy and corticosteroid injections. These second line treatments are important in preventing the need for surgery as a last resort. (6, 7, 8). Corticosteroid injection is an established second line treatment for GTPS that has been shown to be efficacious but not necessarily long term as reported by a randomised study comparing steroid . (9) This notion has been supported by numerous reviews of GTPS management (10, 11, 12, 13). It is therefore imperative to explore treatment options that have the potential for long-lasting benefits, in the form of regenerative medicine are explored. One such is the use of platelet rich plasma (PRP) which will allow regeneration of cells and more robust healing.

   PRP is an autologous blood product which has been postulated to promote healing in damaged or inflamed tissues including muscles, ligaments, bones and tendons. Platelets contain a variety of elements including growth factors and cytokines which are involved in tissue healing. These include platelet derived endothelial growth factor, platelet derived growth factor, transforming growth factor, insulin like growth factor, vascular endothelial growth factor, basic fibroblast growth factor. These growth factors are present in the processes of tissue injury, inflammation and repair. Therefore the theory is the higher the concentration of platelets, the more growth factors there will be present to promote the healing process when administered directly to the area of interest (14). PRP has been applied in other fields of medicine including regenerative therapies in oral and maxillofacial surgery. (15, 16) Over the past decade or so there have been numerous studies of PRP's efficacy in treating inflammatory musculoskeletal conditions similar in pathology to GTPS, such as lateral epicondylitis, patellar tendinitis, rotator cuff pathology, achilles tendonitis and plantar fasciitis. This has been collectively reviewed by several authors with reports of mixed efficacy compared to standard treatments for these conditions with the most promise shown in plantar fasciitis and patellar tendinitis (17, 18). These reviews all report a lack of evidence to fully support or reject PRP's efficacy in these conditions, except for achilles tendonitis where PRP showed no difference compared with placebo in a randomised study (19, 20). PRP's healing or regenerative properties have shown promise in other areas of orthopaedics such as cartilage pathology (14).

   The success of novel regenerative therapy in the form of PRP in a scientifically conducted clinical study will be a major advance in our current knowledge base and will have wider implications for its use in other fields of orthopaedics and will provide better understanding in developing strategies for dealing with similar issues probably even for degenerative conditions.
3. How does the existing literature support this proposal We have completed a systematic literature review which has been submitted for publication. We used NICE healthcare database advanced search (HDAS) via Athens (PubMed, MEDLINE, CINAHL, EMBASE and AMED databases) to conduct our search from their year of inception to October 2017. In total, four studies were included for analysis consisting of two randomised control trials and two case series. We also identified four additional studies from published conference abstracts (one randomised control trial and three case series). 209 patients included in these studies with a mean age ranging from 48 to 76.2 years. Majority were females with three months minimum duration of symptoms. Diagnosis was made using ultrasound or MRI. Included studies used a variety of outcome measures. Improvement was observed during the first 3 months after injection. Significant improvement was also noted when patients were followed up till 12 months post treatment. We found that there is a paucity of evidence reporting the efficacy of PRP in treatment of GTPS. The current literature has revealed that PRP injections are relatively safe and can be effective. Considering the limitations in these studies, we think more large-sample and high-quality randomised clinical trials are required in the future to provide evidence of the efficacy for PRP as a treatment in GTPS.
4. What is the research question / aims and objectives?

   The aim of the trial is to investigate the clinical efficacy of the novel treatment platelet rich plasma (PRP) in treating patients with GTPS. PRP's clinical efficacy will be compared against a placebo injection of normal saline.

   Hypothesis: PRP is an effective treatment for greater trochanteric pain syndrome.
5. Project Plan

Population: Patients with GTPS Intervention: Platelet rich plasma (PRP) injection into trochanteric area under ultrasound guidance Comparator - Placebo of normal saline Outcome: Validated patient reported outcome measures (iHOT-12), Visual Analogue Score for pain (VAS), Modified Harris Hip Score (mHHS) and quality of life outcome (EQ-5D 3L) will be collected at baseline, 3, 6 and 12 months will be compared within and between the PRP and normal saline arms.

Design: The trial will be a two arm single centre double blind randomised control trial. The study will include a two-way comparison between PRP and placebo normal saline injections for treating GTPS. Participants will be reviewed at baseline, 3, 6 and 12 with patient reported outcome measures (PROM) completed at each of these reviews.

Setting: Hospital outpatient Target population: Participants with GTPS will be identified and referred for inclusion in the study by their main care provider (GP, Orthopaedic surgeon, Rheumatologist).

Health technology being assessed: Platelet rich plasma injection (PRP)

Objectives of the Trial :

1. To test the hypothesis that PRP is effective in treating GTPS in patients who have failed conservative management
2. To assess the duration of effect of PRP Outcome Measures Primary: The International Hip Outcome Tool - 12 (iHOT-12) PROM scores Secondary: The Visual Analogue Score for pain (VAS), Modified Harris Hip Score (mHHS) and the EQ-5D 3L scores

Power and sample size:

The primary outcome of interest is the change from baseline to 12 month follow-up for the 12-item International Hip Outcome Tool (iHOT-12). Statistical significance is set at 5% and desired power at 90%, with two tailed tests applied. The minimally clinically important difference (MCID) for the iHOT-12 has been reported as 10 (from 100) and the standard deviation for the change in score from baseline as no greater than 21 by Sansone et al (23). We conservatively assume that change in iHOT score from baseline in the steroid group will be no more than 10 and the change in the iHOT score form baseline in the PRP group will be no less than 27. Using these figures, a minimal sample size at follow up of 66 (33 in each group) will be required. Pilot data obtained by our team suggest that the refusal to participate rate should be no more than 25% and the dropout rate no more than 35% over 12 months. Refusal rates tend to be low in this patient group given the chronic nature of the condition and the fact that patients will only be approached once conservative management has failed. Thus, we will need to approach 135.4 (round up to 136) patients, and recruit 102 patients to achieve our target sample size.

Difference between current and planned care pathway: None

Dissemination Plan:

To ensure that the outputs from the research informs policy and practice and thereby maximises the benefit to patients and the NHS, the following dissemination strategy has been developed using evidence for translating knowledge into practice. From research evidence we know that research is most effectively disseminated using multiple vehicles, ideally with face to face interaction. So, in addition to giving written feedback to study participants, dissemination activities will include development of links with key organisations such as NICE, NHS Information Centre, NHS Commissioning Board and Quality Observatories to contribute to and capitalise on their networks. In addition, media and national and international medical conferences. Furthermore, Publications including Full, Executive Summary and Plain English summary reports of the research, peer review journals and local NHS newsletters and A5 laminate.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Symptoms consistent with GTPS present for at least 6 months
3. Radiological diagnosis of GTPS using MRI, or ultrasound scan if MRI contraindicated
4. Failed conservative management in any other care setting
5. Patient is willing and able to provide written informed consent.

Exclusion Criteria:

1. Lacks capacity to provide consent
2. Has hip joint osteoarthritis requiring treatment on a plain radiograph
3. Presence of confounding pathologies of the hip MRI
4. Any extensive surgery or deformity of the hip on X-ray.
5. Presence of systemic disorders -coagulopathy, active infection, immune system disorders, peripheral neuropathy, malignancy, unresolved fractures.
6. Had any surgical treatment specifically targeted at GTPS e.g. bursectomy/Ilio-tibial band lengthening
7. Pregnancy
8. Anti-coagulant therapy eg warfarin, rivaroxaban, apixaban, dabigatran
9. Haemaglobin <10g/dL or platelets < 150,000/ul
10. Unable to safely stop anti-platelet/NSAID medications eg. Recent cardiac stenting
11. Has lumbar-sacral spine pathology or a recent history of acute hip trauma
12. Has a recent history of acute sciatica
13. Is not able to attend or comply with treatment or follow-up scheduling
14. Participates in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
International Hip Outcome Tool (i-HOT12) | 6 months
  valid and reliable scoring system that assesses patient's ability to return to an active lifestyle through obtaining subjective measures of symptoms, as well as determining emotional and social health status.

SECONDARY OUTCOMES:
Visual analogue score (VAS) | 6 months
  Pain Score uses a scale from 0 (no pain) to 10 (worst pain)
Modified Harris Hip Score (mHHS) | 6 months
  The modified HHS (MHHS) includes pain and function in the assessment. The maximum score of 91 is multiplied by 1.1 to give a total score out of 100.
The 3-level version of EQ-5D (EQ-5D 3L) | 6 months
  descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Malviya, Principal Investigator — Northumbria Healthcare NHS Trust
Locations (1):
- Northumbria Healthcare NHS Trust, Newcastle upon Tyne, TYNE and WEAR, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
this will be discussed with research and development team

REFERENCES:
- [Derived] Oderuth E, Ali M, Atchia I, Malviya A. A double blind randomised control trial investigating the efficacy of platelet rich plasma versus placebo for the treatment of greater trochanteric pain syndrome (the HIPPO trial): a protocol for a randomised clinical trial. Trials. 2018 Sep 21;19(1):517. doi: 10.1186/s13063-018-2907-x. PMID 30241561